CLINICAL TRIAL: NCT02361970
Title: Study on the Role of Gamma Delta T Cells in Sepsis Immunosuppression and Its Molecular Mechanism
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Kang Yan, Director of Intensive Care Unit, West China Hospital
Other Study IDs: Sepsis-kyan0127
Record Dates: First submitted 2015-01-27; First posted 2015-02-12 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Sepsis
Keywords: sepsis; gamma delta T cells; immunosuppression
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood sample was collected to examine extra-cell expression of gamma delta T cells and their intracellular cytokines with or without immuno-stimulants using flow cytometry.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- severe sepsis and septic shock: patients were diagnosed severe sepsis or septic shock
- patient control: Patients after elective surgeries presented with SIRS but without sepsis
- volunteer: Health persons

SUMMARY:
The purpose of the study is to evaluate the status and function of gamma delta T cells in peripheral blood of sepsis patients.

DETAILED DESCRIPTION:
Sepsis therapy is a prominent problem of the modern critical care medicine,and improving the level of sepsis treatment by immune intervention measures is a hot research topic with close attention.Gamma delta T cells is considered as one new T lymphocyte subset in recent years,which playing an important role in resistance to infection,anti-tumor and immune regulating function in the body.First,we played attention to the status and function of gamma delta T cells in peripheral blood of sepsis patients including differentiation marker,subtype and production of related cytokine,and then the molecular mechanism of insufficient gamma delta T cells.At the same time the responsibility of gamma delta T cells of sepsis patients to certain bacteria and viral antigen and the regulation of gamma delta T cells on other natural immune cells including NK cells and mononuclear cells were studied to identify the status and role gamma delta T cells in sepsis immunosuppression by culture in vitro.Further we studied the effect of specific stimulants on proliferation and activation of gamma delta T cells in patients with sepsis and also anti-infection acquired by gamma delta T cells,expecting as an entry point to explore new treatment strategy to sepsis.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms of severe sepsis and septic shock
* age over 18 years

Exclusion Criteria:

* preexisting autoimmune disease
* patients received immuno-suppressive treatment in the previous 6 months
* patients with chronic infection,e.g.tuberculosis,hepatitis or HIV infection,etc.
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICUs of West China Hospital
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The percentage of activated gamma delta T cells | within 24h after recruitment

SECONDARY OUTCOMES:
The percentage of apoptotic gamma delta T cells | within 24h after recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital,Sichuan University, Chengdu, Sichuan, China